CLINICAL TRIAL: NCT05279534
Title: Efficacy and Safety of Lactobacillus Plantarum and Pediococcus Acidilactici as Twice-daily Co-adjuvant Therapy of Upper Respiratory Tract Infections in Children 6 Months to 5 Years Old
Brief Title: Efficacy and Safety of L. Plantarum and P. Acidilactici in Children With Upper Respiratory Tract Infections
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: AB Biotics, SA (Industry)
Collaborators: Innovacion y Desarrollo de Estrategias en Salud (Other); Hospital General Dr. Manuel Gea González (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PROPED-URTI
Record Dates: First submitted 2022-03-07; First posted 2022-03-15 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Upper Respiratory Tract Infections; Pharyngitis; Tonsillitis
Keywords: Probiotic
MeSH Terms: conditions — Respiratory Tract Infections; Pharyngitis; Tonsillitis | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Randomized controlled trials. Study subjects (6 months to 5 years-old) will be allocated to receive a combination of strains Lactobacillus plantarum CECT30292, Lactobacillus plantarum CECT7484, Lactobacillus plantarum CECT7485, and P. acidilactici CECT7483 (arm one) or placebo (arm two)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study staff, including the Principal Investigator and the persons performing the subject assessments, will be blinded during the study. Sealed individual treatment code envelopes will be kept at the clinic to be able to break the code if any emergency occurs, as judged by the Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Active test product contains four lactic acid bacteria strains with Qualified Presumption of Safety (QPS) status by European Food Safety Authority (EFSA): Lactobacillus plantarum CECT30292, Lactobacillus plantarum CECT7484, Lactobacillus plantarum CECT7485, and Pediococcus acidilactici CECT7483, with maltodextrin (E1400, qs) as excipient, formulated in a vegetable hydroxymethylpropyl-cellulose capsule (HPMC) of size 0. Active test product is a food supplement and not an investigational medicinal product
  Interventions: Dietary Supplement: Probiotic
- Control (Placebo Comparator): The control study product is identical in packaging and formulation except that none of strains Lactobacillus plantarum CECT30292, Lactobacillus plantarum CECT7484, Lactobacillus plantarum CECT7485 and Pediococcus acidilactici CECT7483 (probiotic bacteria) are present. The Control product contains maltodextrin (E1400, qs) only, in a vegetable hydroxymethylpropyl-cellulose capsule (HPMC) of size 0.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Combination of strains Lactobacillus plantarum CECT30292, Lactobacillus plantarum CECT7484, Lactobacillus plantarum CECT7485, and Pediococcus acidilactici CECT7483, twice daily for 15 days
  Arms: Probiotic
Other: Placebo — Combination of maltodextrin (E1400, qs) in a vegetable hydroxymethylpropyl-cellulose capsule (HPMC) of size 0, twice daily for 15 days
  Arms: Control

SUMMARY:
Randomized, placebo-controlled trial to evaluate the coadjuvant effect of a combination of L. plantarum and P. acidilactici probiotic strains, taken twice daily, in children 6 months to 5 years-old with upper respiratory tract infections with pharyngitis and/or tonsillitis. Main objective is to evaluate efficacy of this probiotic in reducing fever and pain, as well to evaluate its safety.

DETAILED DESCRIPTION:
Randomized, placebo-controlled trial (RCT) to evaluate the coadjuvant effect of probiotic strains L. plantarum CECT30292, L.plantarum CECT7484 and CECT7485 together with P. acidilactici CECT7483, taken twice daily, in children 6 months to 5 years-old with upper respiratory tract infections with pharyngitis and/or tonsillitis, as diagnosed by a physician.

Main objective is to evaluate efficacy of this probiotic in reducing fever (as per infrared thermometer, same model for all recruited subjects) and pain (as per FLACC scale [Face, Legs, Activity, Cry and Consolability]), as well to evaluate its safety. Secondary objectives include effect on cough, rhinorrhea, nasal congestion, use of concomitant medication, emergency visits, hospitalizations, schooling absences and salivary immune markers.

Probiotic intervention will last 15 days, and patients will return for follow-up visits on the last day of probiotic intervention (day 15), and well as day 30 and 60.

The study aims at enrolling and randomizing 80 children fulfilling entry criteria and living in Mexico City area (2,200m over the sea level), after parents or legal guardians sign informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children, 6 months to 5 years-old
* Diagnosed with upper respiratory tract infection with pharyngitis and/or tonsillitis by a physician
* With fever >37.5 Celsius degrees and FLACC (Face, Legs, Activity, Cry and Consolability) score >3
* Symptom onset no more than 48h before study entry
* Body weight at birth >2500 gr
* Informed consent provided by parents or legal guardians

Exclusion Criteria:

* Failure to thrive
* Asthma or significant allergic disease
* Use of antibiotics, antivirals, probiotics or prebiotics for more than 48h within 2 weeks of study entry
* History of recurrent respiratory infections (>2 otitis, >1 severe sinusitis or >1 pneumonia) within 12 months of study entry
* History of 2 or more invasive infections (meningitis, cellulitis, osteomyelitis, sepsis)
* Chronic diarrhea or short bowel syndrome
* Congenital heart or respiratory deficiency
* Known alpha1-antitrypsin deficiency
* Concurrent participation in other clinical trial(s)
* Other particular conditions which, in the judgment of the Principal Investigator, may interfere with the study

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Daily evolution of fever | Day 1 to 15
  Daily severity of fever (Celsius degrees), as measured with an infrared thermometer (same model for all recruited subjects) and noted in patient diary
Daily evolution of pain | Day 1 to 15
  Daily severity of pain, as per FLACC scale (Face, Legs, Activity, Cry and Consolability, ranging 0 [no pain] to 10 [maximum pain]) and noted in patient diary

SECONDARY OUTCOMES:
Fever Area Under the Curve | Day 1 to 60
  Area Under the Curve (AUC) of daily fever (body temperature, Celsius degrees)
Pain Area Under the Curve | Day 1 to 60
  Area Under the Curve (AUC) of daily pain, as per FLACC scale (Face, Legs, Activity, Cry and Consolability, ranging 0 [no pain] to 10 [maximum pain])
Days with fever | Day 1 to 60
  Days with body temperature > 37.5 Celsius, as noted in patient diary
Days with pain | Day 1 to 60
  Days with pain as per FLACC scale (Face, Legs, Activity, Cry and Consolability), as noted in patient diary
Days with rhinorrhea | Day 1 to 60
  Days with runny nose, as noted in patient diary
Days with cough | Day 1 to 60
  Days of cough, as noted in patient diary
Days with nasal congestion | Day 1 to 60
  Days of nasal congestion, as noted in patient diary
Days with any symptom | Day 1 to 60
  Days with one or more of the following symptom: fever, pain, rhinorrhea, cough or nasal congestion (as noted in patient diary)
Days with concomitant medication | Day 1 to 60
  Days of intake of NSAIDS (non-steroidal anti-inflammatory drugs) and/or antihistamines, as noted in patient diary
Number of children receiving antibiotics | Day 1 to 60
  Number of children receiving antibiotics
Number of hospitalizations | Day 1 to 60
  Number of children being hospitalized related to respiratory tract infection
Number of medical or emergency visits | Day 1 to 60
  Number of medical or emergency visits related to respiratory tract infection
Days of schooling absence | Day 1 to 60
  Days of daycare or kindergarten absence, as noted in patient diary
Change in salivary immune biomarkers | Day 1 to 15
  Change in concentration of Immunoglobulin A (IgA), Tumor Necrosis Factor-alpha (TNFa), Interleukin 1-beta (IL-1b) and Interleukin 10 (IL-10) in saliva samples
Total treatment costs | Day 1 to 60
  Cost of medical and emergency visits, drug treatments (anti-inflammatory drugs, anti-histamines and antibiotics) and schooling absence
Time to fever resolution | Day 1 to 15
  Time to body temperature at or below 37.5 Celsius, as noted in patient diary
Time to pain resolution | Day 1 to 15
  Time to FLACC (Face, Legs, Activity, Cry and Consolability, ranging 0 [no pain] to 10 [maximum pain]) score < 2, as noted in patient diary
Time to complete symptom resolution | Day 1 to 15
  Time to clearance of all of the following symptoms: fever, pain, rhinorrhea, cough and nasal congestion, as noted in patient diary
Time to fever recurrence | Day 15 to 60
  Time to body temperature >37.5 Celsius after initial resolution (see outcome #19), as noted in patient diary
Time to pain recurrence | Day 15 to 60
  Time to FLACC (Face, Legs, Activity, Cry and Consolability, ranging 0 [no pain] to 10 [maximum pain]) score > 3 after initial resolution (see outcome #20), as noted in patient diary
Time to any symptom recurrence | Day 15 to 60
  Time to recurrence of any symptom (fever, pain, rhinorrhea, cough and nasal congestion) after initial complete symptom resolution (see outcome #21), as noted in patient diary
Change in microbiota | Day 1 to 15
  Change in microbiota composition, as determined by 16S gene sequencing

OTHER OUTCOMES:
Etiology of the upper respiratory tract infection at baseline | Day 1
  Identification of the viral or bacterial pathogen responsible for the baseline episode of upper respiratory tract infection by molecular methods
Salivary vitamin D at baseline | Day 1
  Concentration of vitamin D at baseline as measured in saliva sample

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gutierrez-Castrellon, MD, PhD, Principal Investigator — Hospital General Dr. Manuel Gea Gonzalez
Locations (1):
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Mexico DF, Mexico

REFERENCES:
- [Background] Manworren RC, Hynan LS. Clinical validation of FLACC: preverbal patient pain scale. Pediatr Nurs. 2003 Mar-Apr;29(2):140-6. PMID 12723828
- [Background] Gutierrez-Castrellon P, Gandara-Marti T, Abreu Y Abreu AT, Nieto-Rufino CD, Lopez-Orduna E, Jimenez-Escobar I, Jimenez-Gutierrez C, Lopez-Velazquez G, Espadaler-Mazo J. Probiotic improves symptomatic and viral clearance in Covid19 outpatients: a randomized, quadruple-blinded, placebo-controlled trial. Gut Microbes. 2022 Jan-Dec;14(1):2018899. doi: 10.1080/19490976.2021.2018899. PMID 35014600
- [Background] Maya-Barrios A, Lira-Hernandez K, Jimenez-Escobar I, Hernandez L, Ortiz-Hernandez A, Jimenez-Gutierrez C, Lopez-Velazquez G, Gutierrez-Castrellon P. Limosilactobacillus reuteri ATCC PTA 5289 and DSM 17938 as adjuvants to improve evolution of pharyngitis/tonsillitis in children: randomised controlled trial. Benef Microbes. 2021 Apr 12;12(2):137-145. doi: 10.3920/BM2020.0171. Epub 2021 Apr 1. PMID 33789556
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806